CLINICAL TRIAL: NCT01067222
Title: Prospective, Randomized, Double-blind Study, Placebo-controlled, Parallel-group, Multi-center Trial Assessing the Effects of BF2.649 in Treatment of Excessive Daytime Sleepiness in Narcolepsy
Brief Title: Efficacy and Safety Study of BF2.649 in the Treatment of Excessive Daytime Sleepiness in Narcolepsy
Acronym: Harmony1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07-03 / BF2.649; 2008-007866-46 (EudraCT Number)
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Narcolepsy; Excessive Daytime Sleepiness; Cataplexy; Sleep Disorders
Keywords: Narcolepsy; Excessive daytime Sleepiness; Cataplexy; Sleep Disorders; Sleep attacks; Orphan Drug; Pitolisant
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence; Cataplexy; Sleep Wake Disorders | interventions — pitolisant; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BF2.649 (Experimental)
  Interventions: Drug: BF2.649
- Modafinil (Active Comparator)
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BF2.649 — BF2.649 oral capsules at 10 or 20 or 40 mg per day
  Other Names: Pitolisant
  Arms: BF2.649
Drug: Modafinil — Modafinil oral capsules at 100 or 200 or 400 mg per day
  Other Names: Modiodal
  Arms: Modafinil
Drug: Placebo — Placebo oral capsules, 4 capsules per day
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of BF2.649 administered by individual titration in narcoleptic patients with excessive daytime sleepiness (EDS)

DETAILED DESCRIPTION:
BF 2.649, a new experimental drug, significantly decreases, in patient with narcolepsy, the excessive daytime sleepiness (EDS) evaluated by Epworth Sleepiness Scale (ESS), according the results of two previous clinical studies.

The objective of this study is to determine the efficacy and safety of BF2.649 administered by escalating dose (10, 20 or 40 mg/d) in narcoleptic patients with excessive daytime sleepiness versus placebo and Modafinil as assessed by both of objective and subjective measures including ESS, MWT, patients sleep diary.

60 patients with narcolepsy with or without cataplexy will be included.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of narcolepsy with or without cataplexy
* patients need to free of or discontinue psychostimulant medications for at least 14 days,
* patients with severe cataplexy are permitted to remain on their anticataplectic medications at stable doses
* patients must have adequate support to comply with the entire study requirements

Exclusion Criteria:

* Other conditions than Narcolepsy that can be considered as the primary causes of excessive daytime sleepiness
* Patients who are unable or unwilling to temporarily discontinue any no-authorized drugs or substances
* Psychiatric and neurological disorders such as psychosis or dementia, bipolar illness, severe anxiety, clinical depression, history of seizure disorder or other problem that in the investigator's opinion would preclude the patient's participation
* Current or recent history of a substance abuse or dependence disorder including alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | between baseline and at the end of 8 week DB phase

SECONDARY OUTCOMES:
Sleep Diary: Number and duration of diurnal sleep and sleepiness episodes, number of cataplexy attacks | 14 days before randomization and 7 days before each visit
Maintenance of Wakefulness Test (MWT), Test of Sustained Attention to Response Task (SART). | at inclusion and after 8-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassetti, Principal Investigator — Neurocenter (EOC) of Southern Switzerland, Lugano, Switzerland
Locations (1):
- Neurocenter (EOC) of Southern Switzerland, Lugano, Switzerland

REFERENCES:
- [Derived] Meskill GJ, Davis CW, Zarycranski D, Doliba M, Schwartz JC, Dayno JM. Clinical Impact of Pitolisant on Excessive Daytime Sleepiness and Cataplexy in Adults With Narcolepsy: An Analysis of Randomized Placebo-Controlled Trials. CNS Drugs. 2022 Jan;36(1):61-69. doi: 10.1007/s40263-021-00886-x. Epub 2021 Dec 21. PMID 34935103
- [Derived] Watson NF, Davis CW, Zarycranski D, Vaughn B, Dayno JM, Dauvilliers Y, Schwartz JC. Time to Onset of Response to Pitolisant for the Treatment of Excessive Daytime Sleepiness and Cataplexy in Patients With Narcolepsy: An Analysis of Randomized, Placebo-Controlled Trials. CNS Drugs. 2021 Dec;35(12):1303-1315. doi: 10.1007/s40263-021-00866-1. Epub 2021 Nov 25. PMID 34822113
- [Derived] Dauvilliers Y, Bassetti C, Lammers GJ, Arnulf I, Mayer G, Rodenbeck A, Lehert P, Ding CL, Lecomte JM, Schwartz JC; HARMONY I study group. Pitolisant versus placebo or modafinil in patients with narcolepsy: a double-blind, randomised trial. Lancet Neurol. 2013 Nov;12(11):1068-75. doi: 10.1016/S1474-4422(13)70225-4. Epub 2013 Oct 7. PMID 24107292